CLINICAL TRIAL: NCT03197649
Title: Randomized, Prospective, Split Scar Pilot Study to Evaluate the Efficacy of CO2 Laser Phototherapy for Management of Mature Burn Scars
Brief Title: CO2 Laser Phototherapy for Management of Mature Burn Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 950482
Record Dates: First submitted 2017-06-14; First posted 2017-06-23 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Burn Scar

STUDY DESIGN:
Intervention Model Description: The study patient will have one portion of their scar, measuring 5x5 cms (or 50% of the scar, for scars smaller than 5x10 cms) left untreated at the time of the study.
Who Masked: Participant
Masking Description: Participant is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No laser phototherapy treatment
- Laser phototherapy treatment (Experimental): Laser phototherapy treatment administered in OR
  Interventions: Procedure: Laser phototherapy treatment

INTERVENTIONS:
Procedure: Laser phototherapy treatment — Laser phototherapy treatment administered in OR
  Arms: Laser phototherapy treatment

SUMMARY:
Evaluate mature burn scars before and after treatment with CO2 for patients age 3-21 while comparing the treated areas to an untreated control area in the same patient.

DETAILED DESCRIPTION:
Laser phototherapy has gained growing acceptance and popularity for management of burn scars. The most commonly used laser is the Carbon Dioxide (CO2) Laser. At this institution, the investigator has used CO2 for management of Burn Scars since 2012. While the existing literature and the investigator's anecdotal experience thus far has been positive overall, there is no conclusive evidence to support that CO2 does indeed improve the quality of mature burn scars

The primary objective of this study is to evaluate mature burn scars before and after treatment with CO2 for patients age 3-21 while comparing the treated areas to an untreated control area in the same patient.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to 21
* Patients with mature burn scars that are at least two years old from burn injury and that have not previously undergone CO2 laser therapy for scar revision.
* Scars in all body areas with the exception of face, genitals or hands will be considered eligible for the study
* Entry into this study is open to pediatric patients of both genders.
* Entry into this study is open to pediatric patients of all ethnic backgrounds.
* Entry into this study is open to females of childbearing potential with a negative urine or serum pregnancy test

Exclusion Criteria:

* Patients with scars less than 2 years old
* Patients with contraindications to laser treatment (i.e.: active acne infections/ treatment with isotretinoin, active Zoster infection)
* Patients receiving other forms of scar revision therapy such as other laser types, steroid injections, or surgical excisions.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Change in scar assessment evaluation | Prior to initial treatment and no sooner than 3 months following last treatment
  Patient and Observer Scar Assessment Scale

CONTACTS AND LOCATIONS:
Overall Officials: Pirko Maguina, MD, Principal Investigator — UC Davis
Locations (1):
- Shriners Hospitals for Children, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan